CLINICAL TRIAL: NCT01782638
Title: Effect of Deep Brain Stimulation on Gait of Patients With Parkinson's Disease Depending on Electrode Location in Subthalamic Area.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0140; 2011-A00892-39
Record Dates: First submitted 2013-01-21; First posted 2013-02-04 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2013-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep brain stimulation; Gait; Freezing; Electrode placements
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- deep brain stimulation with high frequency (Experimental): The primary purpose of this study is to compare the effect of deep brain stimulation with high frequency vs low frequency on gait of patients whatever the electrodes placement (STN ou Forel fields) and whatever the medication condition (with or without treatment).
  Interventions: Behavioral: deep brain stimulation
- low frequency on gait of patients (Other): The primary purpose of this study is to compare the effect of deep brain stimulation with high frequency vs low frequency on gait of patients whatever the electrodes placement (STN ou Forel fields) and whatever the medication condition (with or without treatment).
  Interventions: Behavioral: deep brain stimulation

INTERVENTIONS:
Behavioral: deep brain stimulation

SUMMARY:
Deep brain stimulation of STN (subthalamic nucleus) at high frequencies generally improved gait in parkinsonian patients. However, sometimes the investigators observed a gait aggravation either with using high voltage and high frequencies, either because of suboptimal placement of electrode inside Forel H2 field. The most frequent hypothesise to explain this gait aggravation is a modulation of the activity of pedunculopontine nucleus due to a diffusion of the electric stimulation current to the fibbers going near STN area.

The primary purpose of this study is to compare the effect of deep brain stimulation with high frequency versus low frequency on gait of patients whatever the electrodes placement (STN ou Forel fields) and whatever the medication condition (with or without treatment).

DETAILED DESCRIPTION:
A randomized, double-blind, parallel-group study 2 groups of patients: 10 patients with electrodes placed in STN and 10 patients with electrodes placed in Forel fields.

1 group of healthy paired-control (n=20).

Patients will be evaluated without and with treatment on two mornings (J0 and J0+1day).

In each condition of treatment, 3 conditions of stimulation were tested: without stimulation; frequency 25Hz, frequency 130 Hz.

Evaluations consist on :

* motor evaluation (UPDRS)
* gait evaluation (to walk on a gait mat)
* Stand-Walk-Sit Test

ELIGIBILITY:
Inclusion Criteria:

* Patients :
* Men or women aged between 45 -85 years
* Patients with an idiopathic Parkinson's disease according to UKPDSBB criteria
* Normal neurologic evaluation (except Parkinson's disease)
* Patient treated with a deep brain stimulation according to the French consensus conference of treatment of Parkinson's disease (Consensus Conference Proceeding, 2000)
* Affiliated to National Health system
* Having given their informed consent

Healthy subject

* Men or women aged between 45 -85 years
* Normal neurologic evaluation
* Affiliated to National Health system
* Having given their informed consent

Exclusion Criteria:

* Patients :
* Patients suffering of an atypical Parkinson syndrome
* Patients with locomotive disorders which can interfere in gait evaluation
* Patients with dementia (MMS <24)
* Under guardianship
* In excluding period for another study
* Person who participate to an other study

Healthy subject

* Subject with locomotive disorders which can interfere in gait evaluation
* Subject with dementia (MMS <24)
* Under guardianship
* In excluding period for another study

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04-23 (Actual); Study Completion 2013-04-23 (Actual)

PRIMARY OUTCOMES:
The step length (expressed in meter) | from day 1 (without L Dopa) to day 2 (with L Dopa)

SECONDARY OUTCOMES:
The gait speed | from day 1 (without L Dopa) to day 2 (with L Dopa)
The step cadence | From day 1 (without L Dopa) to day 2 (with L Dopa)
The number of freezing | from day 1 (without L Dopa) to day 2 (with L Dopa)
The UPDRS score | from day 1 (without L Dopa) to day 2 (with L Dopa)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France